CLINICAL TRIAL: NCT06902077
Title: Carb Control: Low-Carbohydrate Dietary Intervention for Pediatric Patients With Type 2 Diabetes
Brief Title: A Low-Carb Approach to Treat Type 2 Diabetes in Pediatric Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Children's of Alabama (Other)
Responsible Party: Principal Investigator, Ortal Resnick, Fellow- Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300014030; 3130035.000.213130035.31165200 (Other Grant/Funding Number: Fellows Research account)
Record Dates: First submitted 2025-03-07; First posted 2025-03-30 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes
Keywords: Pediatric type 2 diabetes; Type 2 Diabetes; low carb diet; Low-Carbohydrate Dietary
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Diet, Diabetic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low carb diet (Active Comparator): Participants in this group will limit the amount of carbohydrates they eat each day to 50-80 grams.
  This means eating fewer sugars and starches (like bread, pasta, rice, and sweets). Instead, meals will focus on protein, healthy fats, and non-starchy vegetables. Participants will track their food and meet with a dietitian to help them stick to the plan.
  Interventions: Behavioral: low carb diet
- Standard of care (Active Comparator): Participants in this group will follow the current standard diet for managing diabetes. This includes balanced meals with carbohydrates, protein, and fats, based on regular diabetes guidelines.
  Participants will track their food and meet with a dietitian to help them stay on track.
  Interventions: Behavioral: diabetic diet

INTERVENTIONS:
Behavioral: low carb diet — diet based on low carb with max 50-80 grams of carbohydrates daily
  Arms: Low carb diet
Behavioral: diabetic diet — Balanced diet based on standard of care recommendations for type 2 diabetes
  Arms: Standard of care

SUMMARY:
The purpose of this project is to test the effect of a low carb diet compared to standard carb diet among adolescents with T2D over a 24-week period.

DETAILED DESCRIPTION:
Background Type 2 diabetes (T2D) in teenagers is becoming a growing health concern. In the U.S., the number of children and teens diagnosed with T2D nearly doubled between 2002 and 2018. Experts predict that in the next 40 years, the number of young people with T2D could quadruple.

T2D in youth is different from T2D in adults. Teens with T2D have more insulin resistance and their bodies struggle to make enough insulin. Unfortunately, common diabetes medications do not stop the disease from getting worse. Better treatment options for young people with T2D are needed.

T2D happens when the body becomes resistant to insulin and the pancreas struggles to keep up. Diet is a key part of managing T2D, but there are no clear guidelines for the best diet for teens with diabetes.

In adults, low-carbohydrate diets (LCDs) have been shown to:

* Lower blood sugar and improve diabetes control
* Improve insulin function and protect the pancreas
* Reduce the need for diabetes medications
* Help with weight loss, especially in areas of harmful fat like the liver and belly

While LCDs have been well-studied in adults, there is very little research on how they affect adolescents with T2D. A few small studies suggest that reducing carbs may help teens with obesity and fatty liver disease, but we need more evidence to know for sure.

Study Objective This study will test whether a low-carbohydrate diet (LCD) can help improve blood sugar control and insulin function in adolescents with T2D. The investigators will compare it to the standard diet for diabetes care.

How the Study Works

The investigators will conduct a randomized controlled trial (RCT), meaning that participants will be randomly placed into one of two groups:

* Low-Carb Diet (LCD): 50-80 grams of carbohydrates per day
* Standard Diabetes Diet (SCD): A diet based on current guidelines

The study will last 24 weeks (6 months). Participants will keep food records and meet with a dietitian to track their progress.

What The Study Will Measure

The investigators will test whether the low-carb diet helps improve:

* Blood sugar control (measured by HbA1c)
* Insulin function and resistance (measured by an oral glucose tolerance test)
* Weight and fat loss, especially in harmful fat stores
* Triglycerides and cholesterol levels
* Need for diabetes medications

What The Study Expect to Find

The investigators believe that teens who follow a low-carb diet will have:

* Better blood sugar control
* Less insulin resistance
* More weight loss, especially from harmful fat
* Lower triglycerides and better cholesterol levels
* Less need for diabetes medications

This study will help us understand whether reducing carbs is a safe and effective way to improve diabetes in teens.

ELIGIBILITY:
Inclusion Criteria:

* Age 12-18
* Diabetes diagnosis >3 months to ensure stable baseline glycemic control
* HbA1C between 6.5- 8.5%
* BMI >85th percentile
* Negative pancreatic autoantibodies
* Stable dose of anti-diabetic drugs GLP-1, metformin, SGLT-2 inhibitors, for 3 months

Exclusion Criteria:

* Current insulin treatment
* Renal impairment measured as creatinine > 1 mg/dL
* Hepatic dysfunction measured as AST and ALT >100 IU/ml

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | Base line, 3 months, 6 months
  HbA1c levels will be measured to assess long-term glycemic control. Unit of Measure: Percent (%).
Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) | Base line, 3 months, 6 months
  HOMA-IR will be calculated using fasting glucose and insulin values collected at baseline. The formula used is:
  HOMA-IR = (fasting insulin [μU/mL] × fasting glucose [mg/dL]) / 405. This index reflects hepatic insulin resistance.
  Units of Measure: Unitless index
Whole Body Insulin Sensitivity Index (WBISI) | Base line, 3 months, 6 months
  WBISI will be calculated using values from the 2-hour Oral Glucose Tolerance Test (OGTT). The formula is:
  WBISI = 10,000 / √(fasting glucose × fasting insulin × mean OGTT glucose × mean OGTT insulin).
  This index reflects peripheral insulin sensitivity.
  Units of Measure: Unitless index

SECONDARY OUTCOMES:
Change in BMI | Base line, 3 months, 6 months
  Weight and height will be combined to report BMI. Weight in kilograms divided by height in meters squared (kg/m²). Height will be measured using a wall-mounted stadiometer.
  Unit of Measure: kg/m²
Change in blood pressure | Base line, 3 months, 6 months
  Systolic and diastolic blood pressure will be measured in triplicate using an automated oscillometric blood pressure monitor after the participant has been seated quietly for 5 minutes.
  Measurement Tool: Automated oscillometric blood pressure monitor
  Unit of Measure: Millimeters of mercury (mmHg)
Change in lipid profile | Base line, 3 months, 6 months
  Fasting lipid profile will be assessed via venous blood sample. Parameters will include total cholesterol, LDL cholesterol, HDL cholesterol, and triglycerides.
  Unit of Measure: Milligrams per deciliter (mg/dL)
Change in body composition | Base line, 3 months, 6 months
  Body composition will be assessed using a validated bioelectrical impedance analysis (BIA) scale, which estimates fat mass, lean mass, and total body water.
  Measurement Tool: Bioelectrical impedance analysis (BIA) scale
  Unit of Measure: Percent body fat (%) and lean mass (%)

CONTACTS AND LOCATIONS:
Overall Officials: Ortal Resnick, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham/ Children's of Alabama, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No